CLINICAL TRIAL: NCT05524480
Title: Accelerating the Implementation of a Breast and Cervical Cancer Screening and HPV Vaccination Intervention for Under-served Hispanics
Brief Title: Accelerating the Implementation of a Breast and Cervical Cancer Screening and HPV Vaccination Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lara Savas, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-1117
Record Dates: First submitted 2022-08-23; First posted 2022-09-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cancer Prevention
Keywords: Implementation Intervention; Cervical Cancer; Breast Cancer; HPV Vaccination
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Twenty community health centers (CHCs) will be recruited and randomized to either the SEMM-Dissemination and Implementation Assistance arm or the SEMM-Usual Implementation Practice arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salud en Mis Manos - Dissemination and Implementation Assistance (Experimental): The multi-component and multi-faceted implementation strategy SEMM-DIA
  Interventions: Behavioral: Salud en Mis Manos - Dissemination and Implementation Assistance
- Salud en Mis Manos - Usual Implementation Practice (Active Comparator): The SEMM-Usual Implementation Practice arm includes all existing SEMM program materials.
  Interventions: Behavioral: Salud en Mis Manos- Usual Implementation Practice

INTERVENTIONS:
Behavioral: Salud en Mis Manos - Dissemination and Implementation Assistance — The experimental arm will utilize the multi-component and multifaceted implementation strategy, SEMM-DIA. This includes elements like 1) A program orientation session (virtual or in-person), 2) Technical Assistance for implementers, such as SEMM Program Manager/ Coordinator and LHWs, 3) SEMM program materials (including LHW Training curriculum, in-reach/ outreach materials, patient tracking forms), and 4) Virtual community support (Project ECHO series).
  Other Names: SEMM-DIA
  Arms: Salud en Mis Manos - Dissemination and Implementation Assistance
Behavioral: Salud en Mis Manos- Usual Implementation Practice — The control arm will undertake SEMM- Usual Implementation Practice, which includes utilizing all existing SEMM program materials (MOPs, LHW Training Curriculum, etc.) which will be shared with clinic staff in PDF form.
  Other Names: SEMM
  Arms: Salud en Mis Manos - Usual Implementation Practice

SUMMARY:
The proposed study will develop and test an implementation strategy called Salud en Mis Manos-Dissemination and Implementation Assistance (SEMM-DIA) which is an internet-accessible cross-platform that includes additional implementation support strategies to increase the reach, effectiveness, and implementation of an evidence-based breast and cervical cancer screening and HPV vaccination program for Latinas (SEMM).

DETAILED DESCRIPTION:
This study tests a multicomponent and multifaceted implementation strategy, SEMM-DIA and serves as a model for developing other implementation strategies designed to build the capacity of clinic leadership, intervention champions, and LHWs to plan, manage, and deliver SEMM. Investigators will examine the effect of SEMM-DIA program implementation in a randomized group trial comparing the impact of SEMM-DIA vs. SEMM- Usual Implementation Practice on the reach, effectiveness, implementation, and cost-effectiveness of SEMM in safety-net clinics.

ELIGIBILITY:
Inclusion Criteria:

Organization inclusion criteria:

* Clinic or community health center (CHC) with LHWs serving Latina populations.
* Expressed intent to participate in the implementation of SEMM.
* Serve low-income populations with low or no-cost screening and vaccination.
* Provide comprehensive primary health care services.

SEMM Participant Inclusion criteria:

* Latinas who self-identify as Hispanic/Latina.
* Latinas who have at least one unmet breast or cervical cancer prevention need, following Electronic Clinical Quality Measures.
* (1) Latinas aged 21-64 years who have not had a Pap test in the past 3 years, and (2) Latinas aged 30-64 who have not had a HPV test in the past 5 years (CMS eCQM ID: CMS124v9).
* (3) Latinas aged 51-74 years who have not had a mammogram in the past 2 years (CMS eCQM ID: CMS125v9).
* (4) Latinas aged 18-26 years who have not initiated HPV vaccination.

  * Note: Some women will have more than one unmet need (e.g., HPV vaccination and pap test), so they will be included in more than one non-adherent group.

Exclusion Criteria:

Organization exclusion criteria:

- Clinics/Community Health Centers not located in Texas.

SEMM Participant Exclusion criteria:

- Latinas with a prior or current cancer diagnosis due to modified cancer screening surveillance guidelines for cancer survivors.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach is measured by the proportion of women who participate in SEMM education sessions among those that are eligible in the clinic (among all eligible patients) & in the community (the number of participants that receive SEMM education). | 4-month follow up
  Reach will assess several factors: Among eligible women, what number participate in SEMM education sessions?
Reach is measured by the proportion of women who participate in SEMM education sessions among those that are eligible in the clinic (among all eligible patients) & in the community (the number of participants that receive SEMM education). | 8-month follow up
  Reach will assess several factors: Among eligible women, what number participate in SEMM education sessions?
Effectiveness (for screening) as measured by the percentage of women who complete mammogram screening among all eligible patients. | Baseline
  Investigators will assess mammogram completion outcomes using EHR data collection. All participants identified as eligible for a mammogram between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for screening) as measured by the percentage of women who complete mammogram screening among all eligible patients. | 4-month follow-up
  Investigators will assess mammogram completion outcomes using EHR data collection. All participants identified as eligible for a mammogram between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for screening) as measured by the percentage of women who complete mammogram screening among all eligible patients. | 8-month follow-up
  Investigators will assess mammogram completion outcomes using EHR data collection. All participants identified as eligible for a mammogram between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for screening) as measured by the percentage of women who complete cervical cancer screening (Pap or HPV screening test) among all eligible patients. | Baseline
  Investigators will assess Pap completion outcomes using EHR data collection. All participants identified as eligible for a Pap or HPV screening test between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for screening) as measured by the percentage of women who complete cervical cancer screening (Pap or HPV screening test) among all eligible patients. | 4-month follow-up
  Investigators will assess Pap completion outcomes using EHR data collection. All participants identified as eligible for a Pap or HPV screening test between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for screening) as measured by the percentage of women who complete cervical cancer screening (Pap or HPV screening test) among all eligible patients. | 8-month follow-up
  Investigators will assess Pap completion outcomes using EHR data collection. All participants identified as eligible for a Pap or HPV screening test between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for HPV vaccination) as measured by the percentage of female patients who initiate or complete an HPV vaccination among all eligible patients. | Baseline
  Investigators will assess HPV vaccination initiation or completion outcomes using EHR data collection. All participants identified as eligible for an HPV vaccination between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for HPV vaccination) as measured by the percentage of female patients who initiate or complete an HPV vaccination among all eligible patients. | 4-month follow-up
  Investigators will assess HPV vaccination initiation or completion outcomes using EHR data collection. All participants identified as eligible for an HPV vaccination between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
Effectiveness (for HPV vaccination) as measured by the percentage of female patients who initiate or complete an HPV vaccination among all eligible patients. | 8-month follow-up
  Investigators will assess HPV vaccination initiation or completion outcomes using EHR data collection. All participants identified as eligible for an HPV vaccination between program implementation start and end (regardless if identified via in-reach or outreach) will serve as the denominator.
The level of Implementation will be assessed the extent to which SEMM has been carried out per clinic. (1) | 8-month follow-up
  Investigators will assess the level of implementation from baseline to 8-month follow-up using manager assessments.
The level of Implementation will be assessed the extent to which SEMM has been carried out per clinic. (2) | 8-month follow-up
  Investigators will assess the level of implementation from baseline to 8-month follow-up using LHW assessments.
The level of Implementation will be assessed the extent to which SEMM has been carried out per clinic. (3) | 8-month follow-up
  Investigators will assess the level of implementation from baseline to 8-month follow-up using in-depth end-of-study interviews with LHWs.
The level of Implementation will be assessed the extent to which SEMM has been carried out per clinic. (4) | 8-month follow-up
  Investigators will assess the level of implementation from baseline to 8-month follow-up using in-depth end-of-study interviews with managers.
Implementation (fidelity) as measured by the degree to which SEMM program components are implemented by LHWs as prescribed. | 4-month follow-up
  Investigators will assess implementation fidelity using participant tracking forms (completed by LHWs) to understand their level of fidelity associated with implementing the program.
Implementation (fidelity) as measured by the degree to which SEMM program components are implemented by LHWs as prescribed. | 8-month follow-up
  Investigators will assess implementation fidelity using end-of-study in-depth interviews with LHWs to understand their level of fidelity associated with implementing the program.
Implementation dose is described as the average dose of SEMM received by participants/delivered by LHWs (time spent in education sessions). | 4-month follow up
  Investigators will assess implementation dose using SEMM participant tracking forms collected for SEMM participants, which record time spent in education sessions.
Implementation dose is described as the average dose of SEMM received by participants/delivered by LHWs (# of navigation calls). | 4-month follow up
  Investigators will assess implementation dose using SEMM participant tracking forms collected for SEMM participants, which record # of navigation calls needed to overcome barriers to complete needed services (mammogram, Pap/HPV test, and HPV vaccination).
Implementation dose is described as the average dose of SEMM received by participants/delivered by LHWs (time spent in education sessions). | 8-month follow up
  Investigators will assess implementation dose using SEMM participant tracking forms collected for SEMM participants, which record time spent in education sessions.
Implementation dose is described as the average dose of SEMM received by participants/delivered by LHWs (# of navigation calls). | 8-month follow up
  Investigators will assess implementation dose using SEMM participant tracking forms collected for SEMM participants, which record # of navigation calls needed to overcome barriers to complete needed services (mammogram, Pap/HPV test, and HPV vaccination).

SECONDARY OUTCOMES:
Cost effectiveness of SEMM-DIA in community and clinic practice settings | 8-month follow up
  The purpose of the economic analysis is to produce information on the cost-effectiveness of SEMM-DIA in community and clinic practice settings. Investigators will determine the current market value of all ingredients associated with the planning and implementation of the dissemination interventions (from study start to 8-month follow-up), including training and other costs of adapting the intervention to specific sites.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Savas, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Maria E Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No